CLINICAL TRIAL: NCT04895371
Title: The Efficacy of Tele-Physiotherapy in Patients After COVID-19 Hospitalization: The PPTCOVID Study
Brief Title: Tele-Physiotherapy After COVID-19 Hospitalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Javaherian, Principal Investigator, Liver Transplantation Research Center, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 99-2-246-49892
Record Dates: First submitted 2021-05-15; First posted 2021-05-20 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Covid19; Coronavirus Disease 2019
MeSH Terms: conditions — COVID-19 | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The participants will be randomly allocated to Tele-physiotherapy or control groups.
  The sample size was calculated to identify clinically relevant effects on the primary outcome, the distance of six-minute walk test. The calculation was performed using STATA 16 software. Presuming a two-sided significance level (α) of 0.05, the power of 80% (β=0.20) and standard deviation based on the results of a relevant study in COVID-19 survivors which assessed the distance of six-minute walk test. Minimal clinically important difference (MCID) of 54m was reported and considered to be clinically significant. Repeated measurement of ANCOVA was used for the calculation with a baseline and two follow-up measurements (correlation of repeated measurement=0.499). After considering 20% possible participants attrition, It was determined that a sample size of 72 participants would be required to detect a significant change, 36 in each group.
Who Masked: Outcomes Assessor
Masking Description: The assessor will be blinded to the randomization and allocation. The assessor will have not access to patients' medical record. Patients will be also asked to do not explain about their procedure to the assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-physiotherapy group (Experimental): Allocated participants to this group will receive 18 physiotherapy sessions (three sessions per week) during six weeks. in these sessions, physiotherapist will prescribe aerobic, resistive, breathing and functional exercises and airway clearance techniques (if needed) based on result of assessment of patients at the discharge phase. the physiotherapist will use some educational contents for the patient and call him/her to guide the patient about how exercises should be performed (determining frequency, time, intensity and type of exercise). the patient should do exercises until next session and provide a feedback. The patient will be assessed weekly using a pre-designed questionnaire remotely. the progression of interventions will be based on the results of weekly assessment.
  Interventions: Other: Tele-physiotherapy group
- Control group (Active Comparator): Allocated participants to control group will receive one consultation session by the physiotherapist. At this session, patients will be educated about how to perform their daily activities, breathing exercises, walking, using oxygen cylinder and dietary.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Tele-physiotherapy group — Allocated participants to this group will receive 18 physiotherapy sessions (three sessions per week) during six weeks. in these sessions, physiotherapist will prescribe aerobic, resistive, breathing and functional exercises and airway clearance techniques (if needed) based on result of assessment of patients at the discharge phase. the physiotherapist will use some educational contents for the patient and call him/her to guide the patient about how exercises should be performed (determining frequency, time, intensity and type of exercise). the patient should do exercises until next session and provide a feedback. The patient will be assessed weekly using a pre-designed questionnaire remotely. the progression of interventions will be based on the results of weekly assessment.
  Arms: Tele-physiotherapy group
Other: Control group — Allocated participants to control group will receive one consultation session by the physiotherapist. At this session, patients will be educated about how to perform their daily activities, breathing exercises, walking, using oxygen cylinder and dietary.
  Arms: Control group

SUMMARY:
Coronavirus disease 2019 (COVID-19), caused by severe acute respiratory syndrome coronavirus 2 (SARS-Cov-2), is a multisystem infectious disease which has led to a global pandemic.

Tele-medicine is a tool to connect patients and health care professions while maintaining social distancing and restrictions. Tele-physiotherapy is a field of physiotherapy which has the advantage of providing therapy.

Since some months ago, different organizations have started the tele-physiotherapy/tele-rehabilitation program to manage the patients' complications after COVID-19. This research team have developed a tele-rehabilitation guideline for physiotherapists to help them how to use tele-physiotherapy program for patients after COVID-19 hospitalization. The aim of this study is to evaluate the efficacy of tele-physiotherapy program in patients discharged after COVID-19.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19), caused by severe acute respiratory syndrome coronavirus 2 (SARS-Cov-2), is a multisystem infectious disease which has led to a global pandemic.

Due to multisystem nature of this disease, it can cause a variety of early and late complications. New studies have revealed some of the long-term sequelae of this disease, such as neurological injuries, arterial or venous thrombosis, cardiac, brain strokes, etc. which need to be taken into consideration during management of patients. Many COVID-19 survivors who require critical care may also develop psychological, physical and cognitive impairments. These patients may develop various impairments because of hospitalization owing to extended immobilization and many hours bed ridden; these include neuromuscular complications, severe muscle weakness and fatigue, joint stiffness, dysphagia, psychological problems, reduced mobility, low quality of life, frequent falls, and even quadriparesis.

Given impacts of COVID-19 on global health care system, innovative approaches in managing patients are needed. This is the reason that tele-medicine is becoming a trendy title for researchers . Tele-medicine is a tool to connect patients and health care professions while maintaining social distancing and restrictions . Digital health interventions can help provide self-monitoring tools, field updates, exercise protocols, and psychological support. Depending on the funding and facilities provided by the health care system, tele-medicine can be designed and employed in each country uniquely.

Physiotherapy interventions can be also delivered through modern digital communication tools. Tele-physiotherapy is a field of physiotherapy which has the advantage of providing therapy wherever is most convenient for the patient through the use of modern digital communication.

Based on the evidences from other outbreak of viruses in the coronavirus strain epidemics, many of the discharged patients after COVID-19 pneumonia are likely to have residual impairment even some years after hospitalization. Not only discharged COVID-19 patients, but also other members of the society might need physiotherapy in this crisis. Despite this need, social distancing should be taken into account and human lives can't be put in danger. Tele-physiotherapy provides a great opportunity for therapists to communicate with their patients, assess and treat them.

Since some months ago, different organizations have started the tele-physiotherapy/tele-rehabilitation program to manage the patients' complications after COVID-19. This research team have developed a tele-rehabilitation guideline for physiotherapists to help them how to use tele-physiotherapy program for patients after COVID-19 hospitalization. The aim of this study is to evaluate the efficacy of tele-physiotherapy program in patients discharged after COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Discharged patients with Covid-19 pneumonia,
* Having at least one rT-PCR Covid test,
* Duration of hospitalization > 10 days,
* Ability to walk,
* Totally oriented,
* Ability to use smartphone,
* Ability to read and write in Persian.

Exclusion Criteria:

* Having any kind of musculoskeletal disorder causing inability to participate in physiotherapy sessions,
* Severe cardiovascular impairments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-06-12 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
6-Minute Walk Test (6MWT) | Baseline
  6-minute walk test is a sub-maximal test to evaluate the aerobic capacity. The distance which patient can walk during 6 minutes will be measured.
6-Minute Walk Test (6MWT) | After six weeks
  6-minute walk test is a sub-maximal test to evaluate the aerobic capacity. The distance which patient can walk during 6 minutes will be measured.
6-Minute Walk Test (6MWT) | After 10 weeks
  6-minute walk test is a sub-maximal test to evaluate the aerobic capacity. The distance which patient can walk during 6 minutes will be measured.

SECONDARY OUTCOMES:
Five Times Sit to Stand test (5TST) | Baseline
  The five times sit to stand is a test which measures the time for sitting and standing from a chair for five times. it is commonly used to assess strength of lower extremity, transitional movements and falling risks in adults.
Five Times Sit to Stand test (5TST) | After six weeks
  The five times sit to stand is a test which measures the time for sitting and standing from a chair for five times. it is commonly used to assess strength of lower extremity, transitional movements and falling risks in adults.
Five Times Sit to Stand test (5TST) | After 10 weeks
  The five times sit to stand is a test which measures the time for sitting and standing from a chair for five times. it is commonly used to assess strength of lower extremity, transitional movements and falling risks in adults.
Fatigue Severity Scale (FSS) | Baseline
  Fatigue Severity Scale is a short nine statement questionnaire which is used to assess the impact of fatigue on individuals. the questionnaire asks the individuals to rate the level of their fatigue. FSS scores vary from 9 to 63 and higher scores present higher fatigue (worsened).
Fatigue Severity Scale (FSS) | After six weeks
  Fatigue Severity Scale is a short nine statement questionnaire which is used to assess the impact of fatigue on individuals. the questionnaire asks the individuals to rate the level of their fatigue. FSS scores vary from 9 to 63 and higher scores present higher fatigue (worsened).
Fatigue Severity Scale (FSS) | After 10 weeks
  Fatigue Severity Scale is a short nine statement questionnaire which is used to assess the impact of fatigue on individuals. the questionnaire asks the individuals to rate the level of their fatigue. FSS scores vary from 9 to 63 and higher scores present higher fatigue (worsened).
International Physical Activity Questionnaire (IPAQ) | Baseline
  The IPAQ is a 27-item subjective measure of physical activity. This instrument is repetitively used instrument to assess the physical activity. This instrument was developed to assess physical activity in adults aged 18-65 years. The Persian version of IPAQ was translated and cross-cultural adapted by Moghaddam et al. (2012).
International Physical Activity Questionnaire (IPAQ) | After six weeks
  The IPAQ is a 27-item subjective measure of physical activity. This instrument is repetitively used instrument to assess the physical activity. This instrument was developed to assess physical activity in adults aged 18-65 years. The Persian version of IPAQ was translated and cross-cultural adapted by Moghaddam et al. (2012).
International Physical Activity Questionnaire (IPAQ) | After 10 weeks
  The IPAQ is a 27-item subjective measure of physical activity. This instrument is repetitively used instrument to assess the physical activity. This instrument was developed to assess physical activity in adults aged 18-65 years. The Persian version of IPAQ was translated and cross-cultural adapted by Moghaddam et al. (2012).
Level of dyspnea | Baseline
  Level of dyspnea is assessed by modified Borg scale. the patient will report his or her level of dyspnea after 6-minute walk test in range of 0(without dyspnea) to 10(most severe dyspnea).
Level of dyspnea | After six weeks
  Level of dyspnea is assessed by modified Borg scale. the patient will report his or her level of dyspnea after 6-minute walk test in range of 0(without dyspnea) to 10(most severe dyspnea).
Level of dyspnea | After 10 weeks
  Level of dyspnea is assessed by modified Borg scale. the patient will report his or her level of dyspnea after 6-minute walk test in range of 0(without dyspnea) to 10(most severe dyspnea).
Short From-36 | Baseline
  Short Form-36 is a self report instrument which evaluate eight domains of health. it is commonly used as a person or population's quality of life.
Short From-36 | After six weeks
  Short Form-36 is a self report instrument which evaluate eight domains of health. it is commonly used as a person or population's quality of life.
Short From-36 | After 10 weeks
  Short Form-36 is a self report instrument which evaluate eight domains of health. it is commonly used as a person or population's quality of life.
Strength of shoulder abduction muscle group | Baseline
  Strength of shoulder abduction muscle group is assessed by hand held dynamometer and will be presented in kilogram.
Strength of shoulder abduction muscle group | After six weeks
  Strength of shoulder abduction muscle group is assessed by hand held dynamometer and will be presented in kilogram.
Strength of shoulder abduction muscle group | After 10 weeks
  Strength of shoulder abduction muscle group is assessed by hand held dynamometer and will be presented in kilogram.
Strength of hip abduction muscle group | Baseline
  Strength of hip abduction muscle group is assessed by hand held dynamometer and will be presented in kilogram.
Strength of hip abduction muscle group | After six weeks
  Strength of hip abduction muscle group is assessed by hand held dynamometer and will be presented in kilogram.
Strength of hip abduction muscle group | After 10 weeks
  Strength of hip abduction muscle group is assessed by hand held dynamometer and will be presented in kilogram.
Strength of knee extension muscle group | Baseline
  Strength of knee extension muscle group is assessed by hand held dynamometer and will be presented in kilogram.
Strength of knee extension muscle group | After six weeks
  Strength of knee extension muscle group is assessed by hand held dynamometer and will be presented in kilogram.
Strength of knee extension muscle group | After 10 weeks
  Strength of knee extension muscle group is assessed by hand held dynamometer and will be presented in kilogram.
Strength of elbow flexion muscle group | Baseline
  Strength of elbow flexion muscle group is assessed by hand held dynamometer and will be presented in kilogram.
Strength of elbow flexion muscle group | After six weeks
  Strength of elbow flexion muscle group is assessed by hand held dynamometer and will be presented in kilogram.
Strength of elbow flexion muscle group | After 10 weeks
  Strength of elbow flexion muscle group is assessed by hand held dynamometer and will be presented in kilogram.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Javaherian, Ph.D. cand., Principal Investigator — Tehran University of Medical Sciences; Mohsen Nasiri-toosi, MD., Study Director — Tehran University of Medical Sciences; Behrouz Attarbashi Moghadam, Ph.D., Study Director — Tehran University of Medical Sciences
Locations (1):
- Imam Khomeini Hospital Complex, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
All related mentioned data will be available through the principle investigator (Email: Javaherian_m@razi.tums.ac.ir) for researchers who provide a related approved proposal and ethical committee approve to achieve aims. These data will be available with publication date until one year.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Until one year after result publication.
Access Criteria: All researchers who provide a related approved proposal and ethical committee approve to achieve aims.

REFERENCES:
- [Background] Enright PL. The six-minute walk test. Respir Care. 2003 Aug;48(8):783-5. PMID 12890299
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Vasheghani-Farahani A, Tahmasbi M, Asheri H, Ashraf H, Nedjat S, Kordi R. The Persian, last 7-day, long form of the International Physical Activity Questionnaire: translation and validation study. Asian J Sports Med. 2011 Jun;2(2):106-16. doi: 10.5812/asjsm.34781. PMID 22375226
- [Background] Bohannon RW. Sit-to-stand test for measuring performance of lower extremity muscles. Percept Mot Skills. 1995 Feb;80(1):163-6. doi: 10.2466/pms.1995.80.1.163. PMID 7624188
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Azimian M, Farahani AS, Dadkhah A, Fallahpour M, Karimlu M. Fatigue severity scale: the psychometric properties of the persian-version in patients with multiple sclerosis. Res J Biol Sci. 2009;4(9):974-7.
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Montazeri A, Goshtasebi A, Vahdaninia M, Gandek B. The Short Form Health Survey (SF-36): translation and validation study of the Iranian version. Qual Life Res. 2005 Apr;14(3):875-82. doi: 10.1007/s11136-004-1014-5. PMID 16022079
- [Background] Thomas P, Baldwin C, Bissett B, Boden I, Gosselink R, Granger CL, Hodgson C, Jones AY, Kho ME, Moses R, Ntoumenopoulos G, Parry SM, Patman S, van der Lee L. Physiotherapy management for COVID-19 in the acute hospital setting: clinical practice recommendations. J Physiother. 2020 Apr;66(2):73-82. doi: 10.1016/j.jphys.2020.03.011. Epub 2020 Mar 30. PMID 32312646
- [Background] World Health Organization. COVID-19 clinical management: living guidance, 25 January 2021. World Health Organization; 2021.
- [Background] SeyedAlinaghi S, Afsahi AM, MohsseniPour M, Behnezhad F, Salehi MA, Barzegary A, Mirzapour P, Mehraeen E, Dadras O. Late Complications of COVID-19; a Systematic Review of Current Evidence. Arch Acad Emerg Med. 2021 Jan 20;9(1):e14. doi: 10.22037/aaem.v9i1.1058. eCollection 2021. No abstract available. PMID 33681819
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Portnoy J, Waller M, Elliott T. Telemedicine in the Era of COVID-19. J Allergy Clin Immunol Pract. 2020 May;8(5):1489-1491. doi: 10.1016/j.jaip.2020.03.008. Epub 2020 Mar 24. No abstract available. PMID 32220575
- [Background] Salawu A, Green A, Crooks MG, Brixey N, Ross DH, Sivan M. A Proposal for Multidisciplinary Tele-Rehabilitation in the Assessment and Rehabilitation of COVID-19 Survivors. Int J Environ Res Public Health. 2020 Jul 7;17(13):4890. doi: 10.3390/ijerph17134890. PMID 32645876
- [Result] Cortes-Telles A, Lopez-Romero S, Figueroa-Hurtado E, Pou-Aguilar YN, Wong AW, Milne KM, Ryerson CJ, Guenette JA. Pulmonary function and functional capacity in COVID-19 survivors with persistent dyspnoea. Respir Physiol Neurobiol. 2021 Jun;288:103644. doi: 10.1016/j.resp.2021.103644. Epub 2021 Feb 27. PMID 33647535
- [Result] Jenkins SC. 6-Minute walk test in patients with COPD: clinical applications in pulmonary rehabilitation. Physiotherapy. 2007 Sep 1;93(3):175-82.
- [Result] Javaherian M, Shadmehr A, Keshtkar A, Beigmohammadi MT, Dabbaghipour N, Syed A, Attarbashi Moghadam B. Safety and efficacy of pulmonary physiotherapy in hospitalized patients with severe COVID-19 pneumonia (PPTCOVID study): A prospective, randomised, single-blind, controlled trial. PLoS One. 2023 Jan 31;18(1):e0268428. doi: 10.1371/journal.pone.0268428. eCollection 2023. PMID 36719885